CLINICAL TRIAL: NCT04317118
Title: Validating the Ask Suicide-Screening Questions (ASQ) for Youth With Autism Spectrum and Neurodevelopmental Disorders
Brief Title: Ask Suicide-Screening Questions (ASQ) for Youth With Autism Spectrum and Neurodevelopmental Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200066; 20-M-0066
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Suicidal Ideation
Keywords: Suicidal Ideation; Suicide Screening; Death; Children; Adolescents
MeSH Terms: conditions — Suicidal Ideation; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurodevelopmental: Individuals between 8 and 17 years old with neurodevelopmental disorders

SUMMARY:
Background:

Suicide is the second leading cause of death for young people ages 10-24 years. There is no gold standard for evaluating suicidal thoughts and behaviors in young people with autism spectrum disorder (ASD) or other neurodevelopmental disorders (NDD). Also, youth with ASD/NDD are often excluded from many research studies. Because of this, researchers need more data. They want to make sure they are asking the best questions for young people in clinics such as the National Institute of Mental Health (NIMH) clinic. They want to make sure they have the best data to determine if a person is at risk for hurting or killing himself or herself.

Objective:

To develop and assess the efficacy of a suicide screening tool for people with ASD/NDD.

Eligibility:

Youth ages 8 to 17 who are engaged in assessment or treatment at the NIMH for ASD or other NDD

Design:

Participants will fill out 4 questionnaires during a 1-hour meeting with study staff. They will answer questions about how they have been feeling. They will be asked if they think about or plan to hurt or kill themselves. They will also be asked if they have ever thought about it or planned it in the past. Other questions will assess their understanding of death. Participants can take a break if needed.

Parents of the participants will be asked similar questions.

Parents will be informed if their child has current thoughts of suicide.

About 1 week after the initial assessment, parents will be contacted to fill out a follow-up questionnaire. It will take about 10 minutes to complete.

DETAILED DESCRIPTION:
Title:

Validating the Ask Suicide-Screening Questions

(ASQ) for Youth with Autism Spectrum and Neurodevelopmental Disorders

Study Description:<TAB>

Currently, no gold standard is available for evaluating suicidal thoughts and behaviors in individuals with Autism Spectrum Disorder (ASD) or other Neurodevelopmental Disorders (NDD). Moreover, youth with ASD/NDD are often excluded from instrument validation studies. Therefore, there is a paucity of sufficiently adapted and validated clinical suicide risk assessments for use with clients with ASD/NDD.

Objectives:

Primary Objective: The main objective of this study is to develop and assess the efficacy of a suicide screening tool for individuals with ASD/NDD.

Secondary Objectives: To assess the sensitivity/specificity of the ASQ in detecting suicide risk in youth with ASD/NDD by comparing its performance to that of the gold-standard clinician s brief suicide safety assessment, and legacy measures. To test the addition/deletion of candidate items on the sensitivity and specificity of the ASQ in detecting suicide risk in youth with ASD/NDD.

Endpoints:<TAB>

Study participation ends when the study measures are completed if/when the study participant does not screen positive on any of the suicide risk measures. If suicidality is detected, they will be treated clinically for suicidal ideation/behavior according to standard clinical practice.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Participants must be engaged in assessment or treatment in one of the inpatient or outpatient medical health settings from one of the study site hospitals that are part of this protocol.
* Participants must be verbally fluent and have the ability to communicate verbally. This will, in part, be determined by one of the patient s clinicians or trained study staff, who will also be an associate investigator for this study and will already have routine access to information regarding the patient s verbal fluency.
* If the parent/patient expresses interest in participating in a research study, verbal fluency will be further confirmed by asking the parents if the child is verbally fluent (e.g. regularly speaks in sentences), asking the parent if their child will be able to understand and answer the study questions, and by observing the subject as they are explaining the study. The observation will entail taking a verbatim language sample if needed and discussing the decision about whether the child meets this verbal fluency criteria with a study supervisor if needed. The data collectors will be at least high school graduates and over the age of 18 and be trained in assessing fluency level through parent interview and observation. They will also be trained to understand the presentation of individuals with ASD, as well as in how to respond if the child is noncompliant or presents with suicidal thoughts and behaviors.
* Age 8 years to 17.
* English speaking child and parent; may use an Augmentative and Alternative Communication (AAC) device to assist.
* A legal guardian must provide permission and participant must sign an assent document or provide verbal assent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* The parent or the legal guardian is unavailable/unwilling to sign consent.
* The participant will not have prisoner status, e.g. not on probation or house arrest

INCLUSION OF VULNERABLE PARTICIPANTS:

-Children: Children and adolescents with ASD/NDD are the focus of the study due to the lack of suicide risk screening tools available for this general population. Clients who do not speak English will be excluded from the study. Unfortunately, the screening tools that will be utilized in this study are not available at this time in any other languages besides English.

OTHER VULNERABLE POPULATIONS:

The study sites include health clinic or psychiatric units that serve children, adolescents or adults with ASD/NDD. Currently these sites service suicidal individuals and no validated instrument with which to assess these vulnerable individuals.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals in either inpatient or outpatient behavioral health settings or research settings.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Suicide risk | Baseline
  A series of candidate items assessing suicide risk, depression, hopelessness, etc. will be used to assess determine participant's suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (3):
- United States (3):
  - Kennedy Krieger Institute/Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Nationwide Children's Hospital/ Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Horowitz LM, Thurm A, Farmer C, Mazefsky C, Lanzillo E, Bridge JA, Greenbaum R, Pao M, Siegel M; Autism and Developmental Disorders Inpatient Research Collaborative (ADDIRC). Talking About Death or Suicide: Prevalence and Clinical Correlates in Youth with Autism Spectrum Disorder in the Psychiatric Inpatient Setting. J Autism Dev Disord. 2018 Nov;48(11):3702-3710. doi: 10.1007/s10803-017-3180-7. PMID 28624965
- [Background] Horowitz LM, Bridge JA, Teach SJ, Ballard E, Klima J, Rosenstein DL, Wharff EA, Ginnis K, Cannon E, Joshi P, Pao M. Ask Suicide-Screening Questions (ASQ): a brief instrument for the pediatric emergency department. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1170-6. doi: 10.1001/archpediatrics.2012.1276. PMID 23027429
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-M-0066.html